CLINICAL TRIAL: NCT04822324
Title: Effects of Spencer's Muscle Energy Technique Along With Strain Counter Strain in Adhesive Capsulitis.
Brief Title: Spencer's Muscle Energy Technique Along With Strain Counter Strain in Adhesive Capsulitis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/00762 Aimen Iftikhar
Record Dates: First submitted 2021-03-22; First posted 2021-03-30 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Adhesive Capsulitis
Keywords: adhesive capsulitis; spencer muscle energy; strain counterstrain
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spencer Muscle energy technique with conventional Physiotherapy (Experimental): 1. shoulder extension with elbow flexion.
  2. shoulder flexion with elbow extension.
  3. circumduction with compression
  4. circumduction with distraction
  5. shoulder abduction and internal rotation with elbow flexion.
  6. shoulder adduction and external rotation with elbow flexion
  7. stretching tissue and pumping fluids with the arm extended: therapist interlocks his fingertips over the deltoid muscle, patient's hand was placed over the therapist shoulder, and the therapist slowly moved the arm away from the shoulder and released.
  During all the movements patient is asked to use their muscle energy against the slight resistance offered by the therapist for 6-8 sec.
  conventional therapy Joint mobilization
  Exercise therapy:
  Self stretching and strengthening exercises
  Interventions: Other: Spencer Muscle energy technique with conventional Physiotherapy
- Strain counter strain along with conventional Physiotherapy and Spencer Muscle energy technique (Active Comparator): Palpate surrounding and opposing tissues to locate tender point for both shoulder abduction and external rotation.
  Use one or two finger pads to monitor fasciculation and TP. Fine-tune position with rotation. Hold the POC (position of comfort) until fasciculation decreases significantly or ceases.
  Average positions hold time while pressure is 90 s to 3 min. Transient periods of brief tingling, numbness, and temperature changes might occur. Release tissue or joint slowly and reassess.
  Interventions: Other: Strain counter strain along with conventional Physiotherapy and Spencer Muscle energy technique

INTERVENTIONS:
Other: Spencer Muscle energy technique with conventional Physiotherapy — shoulder extension with elbow flexion. shoulder flexion with elbow extension. circumduction with compression circumduction with distraction shoulder abduction and internal rotation with elbow flexion. shoulder adduction and external rotation with elbow flexion stretching tissue and pumping fluids with the arm extended: therapist interlocks his fingertips over the deltoid muscle, patient's hand was placed over the therapist shoulder, and the therapist slowly moved the arm away from the shoulder and released.
  During all the movements patient is asked to use their muscle energy against the slight resistance offered by the therapist for 6-8 sec.
  conventional therapy Joint mobilization
  Exercise therapy:
  Self stretching and strengthening exercises
  Arms: Spencer Muscle energy technique with conventional Physiotherapy
Other: Strain counter strain along with conventional Physiotherapy and Spencer Muscle energy technique — Palpate surrounding and opposing tissues to locate tender point for both shoulder abduction and external rotation.
  Use one or two finger pads to monitor fasciculation and TP. Fine-tune position with rotation. Hold the POC (position of comfort) until fasciculation decreases significantly or ceases.
  Average positions hold time while pressure is 90 s to 3 min. Transient periods of brief tingling, numbness, and temperature changes might occur. Release tissue or joint slowly and reassess.
  Arms: Strain counter strain along with conventional Physiotherapy and Spencer Muscle energy technique

SUMMARY:
Numerous Physiotherapy techniques have been found to be beneficial but there is no consensus on the best treatment approach for speeding up rehabilitation process and rejuvenating functional capacity in patients suffering from Adhesive capsulitis. Spencer Muscle energy technique is found to be effective in treatment of shoulder pathologies. It increases pain free range of motion through stretching the tissues, enhancing lymphatic flow and increasing the joint circulation where as Strain Counter Strain is a technique derived from positional release therapy which uses a pain monitor (trigger points) to find the position of the pain when it is no longer felt at the monitoring point. The purpose of this study is to determine the effects of Spencer Muscle energy technique with and without the employment of Strain Counter Strain on pain, Range of motion and disability in Adhesive capsulitis.

DETAILED DESCRIPTION:
Adhesive shoulder capsulitis or arthrofibrosis commonly known as frozen shoulder, depicts a pathological process in which the body forms excessive scar tissue or adhesions in the capsule around the glenohumeral joint, leading to stiffness, pain and dysfunction. The incidence of adhesive capsulitis in general population is approximately three to five percent and up to twenty percent in patients with diabetes. It is more common in women aged between forty and sixty years and in about twenty-thirty percent of cases it occurs bilaterally. In Pakistan, its precise prevalence is unknown, but in general it ranges from two-five percent. Adhesive capsulitis is classified into two categories: primary which is idiopathic in origin and occur spontaneously without any specific trauma or inciting event and is characterized by painful restriction of all shoulder movements, both active and passive, or Secondary which occurs as a result of some identifiable disorder, such as diabetes mellitus, or due to any inciting event such as cardiac surgery or trauma. There are four stages of frozen shoulder. Stage-one is painful shoulder. Stage - two is "Freezing Stage" with chronic pain and limitation in range of motion. Stage-three is "Frozen Stage" with considerable decreased Range Of Motion and rigid "end feel". Stage-four is "Thawing Phase" with progressive improvement in Range Of Motion. Physiotherapy methods such as active and active assisted exercises, pendular ex's, wand ex's, wall and ladder ex's, capsular stretching ex's and shoulder joint mobilization are often standard exercises in treating frozen shoulder. Electrotherapy modalities such as application of ultrasound, Interferential therapy, short-wave diathermy and LASER are used to relieve pain and promote hyperthermal effect to the tissues.

The Spencer technique is a standardized series of shoulder treatments with broad application in diagnosis, treatment and prognosis. It was developed by Spencer in 1961. This approach is a well-known osteopathic manipulative technique that focuses on mobilization of the glenohumeral and scapulothoracic joints. It is an articulatory technique with seven different procedures, in this technique passive, smooth, rhythmic motion of the shoulder joint is done by the therapist to stretch contracted muscles, ligaments and capsule. Most of the force is applied at the end range of motion. This technique increases pain free range of motion through stretching the tissues, enhancing lymphatic flow and stimulating increased joint circulation.

Positional release technique ( PRT), originally termed strain-counterstain, is a therapeutic technique that uses tender points (TPs) and a position of comfort (POC) to resolve the associated dysfunction. Essentially, Positional release technique is the opposite of stretching. For example, if a patient had a tight, tender area on the calf, if the clinician dorsiflex the foot to stretch the calf in an effort to reduce the tightness and pain. This might lead to muscle guarding and increased pain. Using the same example, a clinician who employs Positional release technique would place the tender point in the position of greatest comfort (plantar flexion), shortening the muscle in an effort to relax the tissues and decrease the tender points. Dr. Lawrence H. Jones, an osteopathic physician, was the first to publish a map of tender point locations and their associated treatment positions. Jones1964 proposed that when a muscle is strained by a sudden unexpected force, its antagonist attempts to stabilize the joint, resulting in a counterstain of the muscle in a resting or shortened position. Before the antagonist is counter strained, gamma neural activity is heightened as a result of its shortened position, making the spindle more sensitive propagating development of restriction, sustained contraction, and tender point development. The application of Positional release technique relaxes the muscle-spindle mechanism, decreasing aberrant gamma and alpha neuronal activity, thereby breaking the sustained contraction. The prevailing theory underlying Positional release technique involve spacing tissues in a relaxed shortened state, or position of comfort , for a period of time (ninety sec) to decrease gamma gain in order to facilitate restoration of normal tissue length and tension.

ELIGIBILITY:
Inclusion Criteria:

* Patients clinically diagnosed with unilateral adhesive capsulitis.
* Patients who had restricted ROM (loss of 25% or greater relative to non-
* involved shoulder in one or multidirectional).
* Stage 2 and 3 of frozen shoulder.
* Diabetic patients diagnosed with frozen shoulder.

Exclusion Criteria:

* A history of major shoulder injury or surgery.
* Other disorders possibly influencing existing shoulder symptoms e.g. cervical neuropathy.
* Paralysis or neurological changes of the affected upper limb.
* Fractures or open wounds;
* Degenerative, inflammatory, or infectious arthritis;
* History of intra-articular injection pain treatment.
* History of osteoporosis or malignancies in shoulder region

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS): | 4 weeks
  Numeric Pain Rating Scale (NPRS) is a11-point scale. The scale is anchored on the left with the phrase ''no pain'' and on the right with the phrase ''worst imaginable pain.'' Patients rate their current level of pain and their worst and least amount of pain in the last 24 hours.
Shoulder Pain and Disability Index (SPADI): | 4 weeks
  Functional Disability was measured using Shoulder pain and Disability Index (SPADI). It was developed to measure the pain and disability associated with shoulder pathology. SPADI is a self administered index consisting of 13 items divided into two subscales i.e. pain and disability.
Shoulder ROM | 4 Weeks
  Shoulder ROM was measured using Goniometer. It is an instrument which measures the available range of motion at a joint. There are different types of goniometers. The type that is most used is the universal standard goniometer, which is either made with plastic or metal tool. It consists of a stationary arm, a movable arm and a fulcrum. It is a reliable tool for measuring shoulder ROM's in degree.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Le HV, Lee SJ, Nazarian A, Rodriguez EK. Adhesive capsulitis of the shoulder: review of pathophysiology and current clinical treatments. Shoulder Elbow. 2017 Apr;9(2):75-84. doi: 10.1177/1758573216676786. Epub 2016 Nov 7. PMID 28405218
- [Background] Manske RC, Prohaska D. Diagnosis and management of adhesive capsulitis. Curr Rev Musculoskelet Med. 2008 Dec;1(3-4):180-9. doi: 10.1007/s12178-008-9031-6. PMID 19468904
- [Background] D'Orsi GM, Via AG, Frizziero A, Oliva F. Treatment of adhesive capsulitis: a review. Muscles Ligaments Tendons J. 2012 Sep 10;2(2):70-8. Print 2012 Apr. PMID 23738277
- [Background] Inayat F, Ali NS, Shahid H, Younus F. Prevalence and Determinants of Frozen Shoulder in Patients with Diabetes: A Single Center Experience from Pakistan. Cureus. 2017 Aug 6;9(8):e1544. doi: 10.7759/cureus.1544. PMID 29018641
- [Background] Doner G, Guven Z, Atalay A, Celiker R. Evalution of Mulligan's technique for adhesive capsulitis of the shoulder. J Rehabil Med. 2013 Jan;45(1):87-91. doi: 10.2340/16501977-1064. PMID 23037929
- [Background] Patriquin DA. The evolution of osteopathic manipulative technique: the Spencer technique. J Am Osteopath Assoc. 1992 Sep;92(9):1134-6, 1139-46. PMID 1429074
- [Background] Patel VD, Eapen C, Ceepee Z, Kamath R. Effect of muscle energy technique with and without strain-counterstrain technique in acute low back pain - A randomized clinical trial. Hong Kong Physiother J. 2018 Jun;38(1):41-51. doi: 10.1142/S1013702518500051. Epub 2018 Apr 4. PMID 30930578
- [Background] Mintken PE, Glynn P, Cleland JA. Psychometric properties of the shortened disabilities of the Arm, Shoulder, and Hand Questionnaire (QuickDASH) and Numeric Pain Rating Scale in patients with shoulder pain. J Shoulder Elbow Surg. 2009 Nov-Dec;18(6):920-6. doi: 10.1016/j.jse.2008.12.015. Epub 2009 Mar 17. PMID 19297202
- [Background] Kolber MJ, Hanney WJ. The reliability and concurrent validity of shoulder mobility measurements using a digital inclinometer and goniometer: a technical report. Int J Sports Phys Ther. 2012 Jun;7(3):306-13. PMID 22666645
- [Background] Roach KE, Budiman-Mak E, Songsiridej N, Lertratanakul Y. Development of a shoulder pain and disability index. Arthritis Care Res. 1991 Dec;4(4):143-9. PMID 11188601